CLINICAL TRIAL: NCT01486082
Title: Usefulness of Antimicrobial Susceptibility in the Eradication of Helicobacter Pylori
Brief Title: Antimicrobial Susceptibility for Helicobacter Pylori Eradication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Donostia (Other)
Responsible Party: Principal Investigator, LUIS BUJANDA, Director, Head of Gastroenterology Department, principal investigator, clinical proffesor, Hospital Donostia
Other Study IDs: HP02
Record Dates: First submitted 2011-11-19; First posted 2011-12-06 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: OCA 10; Antibiogram; Eradication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Empirical OCA: This group will be treated with omeprazole, amoxicillin and clarithromycin without having a previous antibiogram.
  Interventions: Other: OCA 10
- OCA after antibiogram: This group will be treated with omeprazole, clarithromycin and amoxicillin after an antibiotic susceptibility confirmation.
  Interventions: Other: OCA 10

INTERVENTIONS:
Other: OCA 10 — A group will be treated with omeprazole (20 mg / 12 h), amoxicillin (1 g/ 12 h)and clarithromycin (500 mg/12 h) for 10 days (as following current guides) without having a previous antibiogram, and the other group will be treated after antibiotic susceptibility.
  Other Names: O: Omeprazole; C: Clarithromycin; A: Amoxicillin

SUMMARY:
Due to the high rate of resistance to clarithromycin in our area the investigators proposed an study to assess the need of antibiogram previous to the empirical OCA 10 treatment, in order to improve the rate of eradication.

DETAILED DESCRIPTION:
Usefulness of antimicrobial susceptibility in the eradication of Helicobacter pylori

PURPOSE

Background:

* The rate of eradication of Helicobacter pylori with standard triple therapy (OCA: omeprazole + clarithromycin + amoxicillin) in our area is less than the expected according to the III Maastricht III consensus. However, the current guidelines recommend the use of this therapy.
* According to the Maastricht III consensus, in populations with high rates of clarithromycin resistance (15-20%) another therapy should be considered, or alternatively, testing antimicrobial susceptibility of the H. pylori prior to treatment.

Objectives:

* To clarify the real rate of eradication with OCA therapy with and without antimicrobial susceptibility in our area (with high rate of resistance to clarythromycin).
* To study which is the diagnostic-therapeutic strategy more cost-effective for the treatment of H. pylori.

Design:

* Participants will be screened with a full medical history.
* Participants will aleatory receive OCA therapy empirically, or after antimicrobial susceptibility test if there is no resistance to clarythromycin, for ten days.
* In all cases the eradication of H. pylori will be checked by 13C urea breath test (UBT) in 8 weeks after the therapy have been finished.
* All the adverse event of the therapy will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of H. pylori infection provided by culture, histology or UBT.
* Patients need and indication to treat (peptic ulcer disease, firs-degree family history of gastric cancer, MALT lymphoma or dyspeptic symptoms)
* Patients must be 18 years or older.

Exclusion criteria:

* Previous treatment for H. pylori eradication.
* Patients who have severe concomitant disease.
* Patients who have previous gastric surgery.
* Patients who have intolerance to any antimicrobial drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators recruited patients who are diagnosed with helicobacter pylori infection in our hospital (Hospital Donostia) or in any of the specialist care centres under the management of the Hospital Donostia.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients in whom Helicobacter pylori was eradicated. | 9 months
  The investigators will measure the rate of eradication in each gruop after OCA treatment. One group receive OCA without antibiogram and the other one after checking the sensitivity to clarithromycin.

SECONDARY OUTCOMES:
Number of patient with adverse event | 9 months
Cost of the eradication of Helicobacter Pylori in each group. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: LUIS BUJANDA, Study Director
Locations (1):
- Hospital Donostia, Donostia / San Sebastian, Guipuzcoa, Spain

REFERENCES:
- [Derived] Martos M, Bujanda L, Salicio Y, Sarasqueta C, Ibarra B, Mendarte U, Fernandez-Reyes M, Cosme A. Clarithromycin for first-line treatment of Helicobacter pylori infection after culture in high-resistance regions. Eur J Gastroenterol Hepatol. 2014 Dec;26(12):1380-4. doi: 10.1097/MEG.0000000000000197. PMID 25229983